CLINICAL TRIAL: NCT04550078
Title: The Postprandial Calcium Absorption of a Milk Derived Calcium Permeate - A Randomized Controlled Cross-over Meal Study
Brief Title: The Postprandial Calcium Absorption of a Milk Derived Calcium Permeate - RENEW Acute Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inge Tetens (Other)
Collaborators: Zealand University Hospital (Other); Arla Foods (Industry); University of Aarhus (Other); Innovation Fund Denmark (Individual)
Responsible Party: Sponsor-Investigator, Inge Tetens, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: M235
Record Dates: First submitted 2020-08-10; First posted 2020-09-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium Carbonate (Active Comparator): 800 mg calcium as calcium carbonate in capsules consumed orally once with a standardized meal.
  Interventions: Dietary Supplement: Calcium Carbonate
- Calcium-enriched permeate (Experimental): 800 mg calcium as calcium permeate in capsules consumed orally once with a standardized meal.
  Interventions: Dietary Supplement: Calcium Permeate
- Maltodextrin (Placebo Comparator): 0 mg calcium as placebo capsules with maltodextrin consumed orally once with a standardized meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Calcium Carbonate — Subjects receive a single-dose of 800 mg calcium as calcium carbonate provided in 6 capsules with a standardized breakfast served in the morning.
  Arms: Calcium Carbonate
Dietary Supplement: Calcium Permeate — Subjects receive a single-dose of 800 mg milk calcium as calcium permeate provided in 6 capsules with a standardized breakfast served in the morning.
  Other Names: Capolac
  Arms: Calcium-enriched permeate
Dietary Supplement: Placebo — Subjects receive a single-dose of 0 mg calcium as placebo with maltodextrin provided in 6 capsules with a standardized breakfast served in the morning.
  Arms: Maltodextrin

SUMMARY:
This is a randomized controlled cross-over meal study with the overall aim to investigate the postprandial calcium absorption from calcium permeate compared with calcium carbonate. The hypothesis is that the bioavailability of calcium permeate is equal to or higher than calcium carbonate. This will be investigated in a cross-over design with 10 postmenopausal women age 50-65 as subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >50 years and <65 years of age by the time of inclusion.
* Subject has been menopausal for 2-5 years.
* Subject willing and able to meet at University Hospital, Køge for three whole days in one month.
* Subject is non-smoking or able not to smoke during clinic visits.
* Subject with no history of osteoporotic fractures.
* Subject is willing and able to provide written informed consent prior to participation.

Exclusion Criteria:

* Subject taking supplements or medicine that affects calcium and bone metabolism e.g. diuretics or hormone replacement therapy.
* Subject with vitamin D insufficiency defined as ≤50nmol/l.
* Subject with an osteoporosis diagnosis.
* Presence of renal, gastrointestinal, hepatic or endocrinological diseases.
* Subject with any serious illness e.g. cancer.
* Subject with lactose intolerance.
* Subject with celiac disease.
* Known or suspected abuse of alcohol or recreational drugs.
* Known or suspected hypersensitivity to trial products or related products.
* Subject where it is not possible to obtain sufficient data.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Serum Ionized calcium concentration | 3 months
  Blood samples are collected 5 times during subjects three visits. At each visit one baseline measurement blood sample will be collected, followed by measurement 60 minutes, 120 minutes, 240 minutes and 360 minutes after ingestion of study products (calcium carbonate, calcium permeat or placebo).

SECONDARY OUTCOMES:
Serum calcium concentration | 3 months
  Blood samples are collected 5 times during subjects three visits. At each visit one baseline measurement blood sample is collected, followed by measurement 60 minutes, 120 minutes, 240 minutes and 360 minutes after ingestion of study products (calcium carbonate, calcium permeat or placebo).
Serum phosphate concentration | 3 months
  Blood samples are collected 5 times during subjects three visits. At each visit one baseline measurement blood sample is collected, followed by measurement 60 minutes, 120 minutes, 240 minutes and 360 minutes after ingestion of study products (calcium carbonate, calcium permeat or placebo).
Serum magnesium concentration | 3 months
  Blood samples are collected 5 times during subjects three visits. At each visit one baseline measurement blood sample is collected, followed by measurement 60 minutes, 120 minutes, 240 minutes and 360 minutes after ingestion of study products (calcium carbonate, calcium permeat or placebo).
Serum PTH concentration | 3 months
  Blood samples are collected 5 times during subjects three visits. At each visit one baseline measurement blood sample is collected, followed by measurement 60 minutes, 120 minutes, 240 minutes and 360 minutes after ingestion of study products (calcium carbonate, calcium permeat or placebo).
Urinary calcium concentration | 3 months
  Subjects are instructed in 24 hour urine collection for each visit. On visit days two spot-urine samples will be sent for analysis. Samples will be collected at baseline and 360 minutes after ingestion of study products (calcium carbonate, calcium permeate and placebo)
Urine phosphate concentration | 3 months
  Subjects are instructed in 24 hour urine collection for each visit. On visit days two spot-urine samples will be sent for analysis. Samples will be collected at baseline and 360 minutes after ingestion of study products (calcium carbonate, calcium permeate and placebo)
Urine magnesium concentration | 3 months
  Subjects are instructed in 24 hour urine collection for each visit. On visit days two spot-urine samples will be sent for analysis. Samples will be collected at baseline and 360 minutes after ingestion of study products (calcium carbonate, calcium permeate and placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Tetens, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No